CLINICAL TRIAL: NCT03237234
Title: SCIMS Project 1: Enhancing Corticospinal Activation for Improved Walking Function
Brief Title: Enhancing Corticospinal Activation for Improved Walking Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Edelle Field-Fote, PT, PhD, Director of Spinal Cord Injury Research, Shepherd Center, Atlanta GA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCIMS1-703
Record Dates: First submitted 2017-07-13; First posted 2017-08-02 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Motor Training + Sham tDCS (Sham Comparator): Individuals will participate in 3 consecutive sessions of lower extremity motor skill training while receiving sham transcranial direct current stimulation (tDCS).
  Interventions: Other: Motor Skill Training
- Motor Training + tDCS (Experimental): Individuals will participate in 3 consecutive sessions of lower extremity motor skill training combined with transcranial direct current stimulation (tDCS) delivered at 2mA to the motor cortex.
  Interventions: Other: Motor Skill Training; Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Other: Motor Skill Training — Motor skill training will consist of activities that will be performed while standing to promote upright control (the toe-tapping activity will be performed while seated). Participants will perform each of the 6 different activities for one minute each, until 4 cycles of the circuit have been completed (approximately 25 minutes total). Motor training activities will be performed at an intensity of 40-59% of heart rate reserve (HRR). Toe tapping will provide the opportunity for scheduled rest. During MT, all participants will wear a heart rate monitor to ensure that the optimal HR range is achieved. HRR will be calculated from resting and peak heart rate measures obtained during baseline testing via administration of a graded-exercise test.
Device: Transcranial direct current stimulation (tDCS) — The tDCS electrode placement is based on procedures shown to improve gait and balance in a single session when used in combination with gait training activities. tDCS electrodes can simultaneously activate the bilateral leg motor areas when placed at the midline of the scalp slightly anterior to the vertex (anode) and at the inion (cathode), with a current intensity of 2mA. The tDCS device is lightweight, and can be worn in a backpack during the MT activities. As reported previously, participants in the MT-only group will receive sham tDCS to maintain analogous study procedures.
  Arms: Motor Training + tDCS

SUMMARY:
For many people with spinal cord injury (SCI), the goal of walking is a high priority. There are many approaches available to restore walking function after SCI; however, these approaches often involve extensive rehabilitation training and access to facilities, qualified staff, and advanced technology that make practicing walking at home difficult. For this reason, developing training approaches that could be easily performed in the home would be of great value. In addition, non-invasive brain stimulation has the potential to increase the effectiveness of communication between the brain and spinal cord. Combining motor skill training with brain stimulation may further enhance the restoration of function in persons with SCI. Based on these findings, the primary aim of this proof-of-concept study is to inform future intervention development. To meet this aim, we will determine if moderate-intensity, motor skill training can improve walking-related outcomes among persons with SCI and to determine if the addition of non-invasive brain stimulation will result in greater improvements in function compared to training alone.

DETAILED DESCRIPTION:
For many people with spinal cord injury (SCI), the goal of walking is a high priority. There are many approaches available to restore walking function after SCI; however, these approaches often involve access to intensive training programs, facilities, qualified staff, and advanced technology that make practicing walking at home difficult. For this reason, developing training approaches that could be easily performed in the home would be of great value. In addition, research suggests that enhancing brain excitability might have benefits for improving the communication between the brain and spinal cord. Transcranial direct current stimulation (tDCS) is a type of non-invasive brain stimulation that has been shown to directly increase brain excitability, which may make it easier for the brain and nervous system to respond to training. Combining motor skill exercises with brain stimulation may enhance the restoration of walking function in persons with SCI. Based on these findings, the primary aim of this proof-of-concept study is to inform future intervention development. To meet this aim, we will determine if moderate-intensity, motor skill training can improve walking-related outcomes among persons with SCI and to determine if the addition of non-invasive brain stimulation will result in greater improvements in function compared to training alone.

Participants in the proposed study will complete one baseline testing session, 3 motor training sessions, and one follow-up session over 5 consecutive days. During the first and fifth sessions, participants will complete assessments only, which will take approximately 2-3 hours each day. During the second, third, and fourth sessions, participants will perform a series of 6 standing motor skill exercises designed to challenge balance, lower extremity coordination, agility, and speed. Participants will be randomized to either a motor training only group or a motor training + tDCS group. The motor training + tDCS group will receive brain stimulation during the motor skill training, while the motor training only group will receive sensory level brain stimulation only. Each participant will complete the 6 motor skill exercise circuit 4 times. Motor training exercise sessions will last approximately 25-30 minutes and will be preceded and followed by assessments of walking function, spasticity, and ankle strength in order to determine changes in these measures over time.

ELIGIBILITY:
Inclusion Criteria:

* Have a spinal cord injury (neurological level C3-T10);
* Chronic SCI (12 months or greater);
* Neurological impairment classification C or D;
* Able to stand for at least 5 minutes (with or without an assistive device);
* Able to move each leg independently for at least 3 steps;
* Able to rise from sit to stand with moderate assistance from one person;
* Ability and willingness to consent and authorize use of personal health information.

Exclusion Criteria:

* Progressive spinal lesions including degenerative, or progressive vascular disorders of the spine and/or spinal cord;
* Injuries below the neurological spinal level of T10;
* History of cardiovascular irregularities;
* Altered cognitive status;
* Presence of orthopedic conditions that would adversely affect participation in exercise;
* Implanted metallic objects in the head;
* History of seizures;
* Inability and unwillingness to consent and authorize use of personal health information.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Shepherd Center, Inc., Atlanta, Georgia, United States

REFERENCES:
- [Derived] Evans NH, Suri C, Field-Fote EC. Walking and Balance Outcomes Are Improved Following Brief Intensive Locomotor Skill Training but Are Not Augmented by Transcranial Direct Current Stimulation in Persons With Chronic Spinal Cord Injury. Front Hum Neurosci. 2022 May 11;16:849297. doi: 10.3389/fnhum.2022.849297. eCollection 2022. PMID 35634208
- [Derived] Evans NH, Field-Fote EC. A Pilot Study of Intensive Locomotor-Related Skill Training and Transcranial Direct Current Stimulation in Chronic Spinal Cord Injury. J Neurol Phys Ther. 2022 Oct 1;46(4):281-292. doi: 10.1097/NPT.0000000000000403. Epub 2022 May 11. PMID 35544283

RESULTS

PARTICIPANT FLOW:
Groups:
- Motor Skill Training + Sham tDCS (MST+Sham-tDCS): Individuals will participate in 3 consecutive sessions of lower extremity motor skill training while receiving sham transcranial direct current stimulation (MST+sham-tDCS).
  Motor Skill Training: Motor skill training will consist of activities that will be performed while standing to promote upright control (the toe-tapping activity will be performed while seated). Participants will perform each of the 6 different activities for one minute each, until 4 cycles of the circuit have been completed (approximately 25 minutes total). Motor training activities will be performed at an intensity of 40-59% of heart rate reserve (HRR). Toe tapping will provide the opportunity for scheduled rest. During MT, all participants will wear a heart rate monitor to ensure that the optimal HR range is achieved. HRR will be calculated from resting and peak heart rate measures obtained during baseline testing via administration of a graded-exercise test.
- Motor Skill Training + tDCS (MST+tDCS): Individuals will participate in 3 consecutive sessions of lower extremity motor skill training combined with transcranial direct current stimulation (MST+tDCS) delivered at 2mA to the motor cortex.
  MST: Motor skill training will consist of activities performed while standing to promote upright control (the toe-tapping activity will be performed while seated). Participants will perform each of the 6 different activities for one minute each, until 4 cycles of the circuit have been completed (approximately 25 minutes total). Motor training activities will be performed at an intensity of 40-59% of heart rate reserve (HRR). Toe tapping will provide the opportunity for scheduled rest. During MST, all participants will wear a heart rate monitor to ensure that the optimal HR range is achieved. HRR will be calculated from resting and peak heart rate measures obtained during baseline testing via administration of a graded-exercise test.
  Transcranial direct current stimulation (tDCS): The tDCS electrode placement is based on procedures shown to improve gait and balance in a single session when used in combination with gait training activities. tDCS electrodes can simultaneously activate the bilateral leg motor areas when placed at the midline of the scalp slightly anterior to the vertex (anode) and at the inion (cathode), with a current intensity of 2mA.
Period: Overall Study
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Motor Skill Training + Sham tDCS (MST+Sham-tDCS): Individuals will participate in 3 consecutive sessions of lower extremity motor skill training while receiving sham transcranial direct current stimulation (sham-tDCS).
  MST: Motor skill training will consist of activities that will be performed while standing to promote upright control (the toe-tapping activity will be performed while seated). Participants will perform each of the 6 different activities for one minute each, until 4 cycles of the circuit have been completed (approximately 25 minutes total). Motor training activities will be performed at an intensity of 40-59% of heart rate reserve (HRR). Toe tapping will provide the opportunity for scheduled rest. During MST, all participants will wear a heart rate monitor to ensure that the optimal HR range is achieved. HRR will be calculated from resting and peak heart rate measures obtained during baseline testing via administration of a graded-exercise test.
- Motor Skill Training + tDCS (MST+tDCS): Individuals will participate in 3 consecutive sessions of lower extremity motor skill training combined with transcranial direct current stimulation (tDCS) delivered at 2mA to the motor cortex.
  MST: Motor skill training will consist of activities that will be performed while standing to promote upright control (the toe-tapping activity will be performed while seated). Participants will perform each of the 6 different activities for one minute each, until 4 cycles of the circuit have been completed (approximately 25 minutes total). Motor training activities will be performed at an intensity of 40-59% of heart rate reserve (HRR). Toe tapping will provide the opportunity for scheduled rest. During MST, all participants will wear a heart rate monitor to ensure that the optimal HR range is achieved. HRR will be calculated from resting and peak heart rate measures obtained during baseline testing via administration of a graded-exercise test.
  Transcranial direct current stimulation (tDCS): The tDCS electrode placement is based on procedures shown to improve gait and balance in a single session when used in combination with gait training activities. tDCS electrodes can simultaneously activate the bilateral leg motor areas when placed at the midline of the scalp slightly anterior to the vertex (anode) and at the inion (cathode), with a current intensity of 2mA. The tDCS device is lightweight, and can be worn in a backpack during the MST activities.
- Total: Total of all reporting groups
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS) | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (15) | 50.5 (10.7) | 48.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 10 | 8 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 25
10 Meter Walk Test (walk speed) [Mean (Standard Deviation); unit: m/sec] | 0.72 (0.53) | 0.64 (0.51) | 0.69 (0.51)
Spatiotemporal Gait Characteristic (Cadence) [Mean (Standard Deviation); unit: strides/min] | 73.9 (34.3) | 70.7 (38.5) | 72.5 (35.5)
Spatiotemporal Gait Characteristic (symmetry index) [Mean (Standard Deviation); unit: Absolute %] | 14.6 (12.2) | 12.3 (7.4) | 13.6 (10.2)
Spatiotemporal Gait Characteristic (stride length -weaker limb) [Mean (Standard Deviation); unit: cm] | 106.6 (33.5) | 95.0 (33.4) | 101.5 (33.3)
Spatiotemporal Gait Characteristic (stride length - stronger limb) [Mean (Standard Deviation); unit: cm] | 106.8 (33.1) | 94.4 (32.9) | 101.3 (33.0)
Ankle Dorsiflexor Strength (MVC force) [Mean (Standard Deviation); unit: lbs] | 61.9 (35.3) | 66.1 (19.9) | 63.8 (29.0)

OUTCOME MEASURES:

1. Primary Outcome: 10 Meter Walk Test (Walk Speed)
Description: Walking speed was the primary outcome measure for walking function, as speed has been the standard measure used in the literature and allowed us to assess outcomes relative to other published studies. Walking speed was determined using the 10-Meter Walk Test. Participants completed 3 walk trials at each time point, separated by 2 minutes of seated rest. The average walking speed of 3 walks was calculated and used in the analyses. Data reported were obtained at baseline at Day 1 (D1) and at follow-up on Day 5 (D5), 24-hours post-intervention.
Time Frame: D1, D5
Measure: Mean (Standard Deviation); unit: m/sec
Groups:
- Motor Skill Training + Sham tDCS (MST+Sham-tDCS): Individuals will participate in 3 consecutive sessions of lower extremity motor skill training while receiving sham transcranial direct current stimulation (MST+sham-tDCS).
  Motor Skill Training: Motor skill training will consist of activities that will be performed while standing to promote upright control (the toe-tapping activity will be performed while seated). Participants will perform each of the 6 different activities for one minute each, until 4 cycles of the circuit have been completed (approximately 25 minutes total). Motor training activities will be performed at an intensity of 40-59% of heart rate reserve (HRR). Toe tapping will provide the opportunity for scheduled rest. During MST, all participants will wear a heart rate monitor to ensure that the optimal HR range is achieved. HRR will be calculated from resting and peak heart rate measures obtained during baseline testing via administration of a graded-exercise test.
- Motor Skill Training + tDCS (MST+tDCS): Individuals will participate in 3 consecutive sessions of lower extremity motor skill training combined with transcranial direct current stimulation (MST+tDCS) delivered at 2mA to the motor cortex.
  Motor Skill Training: Motor skill training will consist of activities that will be performed while standing to promote upright control (the toe-tapping activity will be performed while seated). Participants will perform each of the 6 different activities for one minute each, until 4 cycles of the circuit have been completed (approximately 25 minutes total). Motor training activities will be performed at an intensity of 40-59% of heart rate reserve (HRR). Toe tapping will provide the opportunity for scheduled rest. During MST, all participants will wear a heart rate monitor to ensure that the optimal HR range is achieved. HRR will be calculated from resting and peak heart rate measures obtained during baseline testing via administration of a graded-exercise test.
  Transcranial direct current stimulation (tDCS): The tDCS electrode placement is based on procedures shown to improve gait and balance in a single session when used in combination with gait training activities. tDCS electrodes can simultaneously activate the bilateral leg motor areas when placed at the midline of the scalp slightly anterior to the vertex (anode) and at the inion (cathode), with a current intensity of 2mA. The tDCS device is lightweight, and can be worn in a backpack during the MST activities.
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
m/sec
  Day 1 (D1) | 0.72 (0.53) | 0.64 (0.51)
  Day 5 (D5) | 0.85 (0.56) | 0.78 (0.46)

2. Secondary Outcome: Spatiotemporal Gait Characteristic (Cadence)
Description: Gait quality was quantified by spatiotemporal gait characteristics (cadence [strides/min], stride length [cm] and step length [cm] of the weaker and stronger limbs) collected via instrumented walkway (GAITRite, CIR Systems Inc., NJ, USA) as participants completed three, 10-Meter Walk Test trials at each time point. Cadence for each walk trial was computed using the GAITRite system, and the average cadence across three walks was used in the analyses. Results are reported for data obtained at baseline Day-1 (D1) and at follow-up on Day-5, 24-hours post-intervention.
Time Frame: D1, D5
Measure: Mean (Standard Deviation); unit: strides/min
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
strides/min
  Day 1 (D1) | 73.9 (34.3) | 70.7 (38.5)
  Day 5 (D5) | 81.5 (34.9) | 82.1 (34.9)

3. Secondary Outcome: Spatiotemporal Gait Characteristic (Stride Length - Weaker Limb)
Description: Gait quality was quantified by spatiotemporal gait characteristics (cadence [strides/min], stride length [cm] and step length [cm] of the weaker and stronger limbs) collected via instrumented walkway (GAITRite, CIR Systems Inc., NJ, USA) as participants completed three, 10-Meter Walk Test trials at each time point. Average stride length of the weaker limb for each walk trial was computed from data obtained from the GAITRite system, and the average stride length across three walks was used in the analyses. Results are reported for data obtained at baseline Day-1 (D1) and at follow-up on Day-5, 24-hours post-intervention.
Time Frame: D1, D5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
cm
  Day 1 (D1) | 106.6 (33.5) | 95.0 (33.4)
  Day 5 (D5) | 114.7 (35.6) | 104.5 (27.8)

4. Secondary Outcome: Spatiotemporal Gait Characteristic (Stride Length - Stronger Limb)
Description: Gait quality was quantified by spatiotemporal gait characteristics (cadence [strides/min], stride length [cm] and step length [cm] of the weaker and stronger limbs) collected via instrumented walkway (GAITRite, CIR Systems Inc., NJ, USA) as participants completed three, 10-Meter Walk Test trials at each time point. Average stride length of the stronger limb for each walk trial was computed from data obtained from the GAITRite system, and the average stride length across three walks was used in the analyses. Results are reported for data obtained at baseline Day-1 (D1) and at follow-up on Day-5, 24-hours post-intervention.
Time Frame: D1, D5
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
cm
  Day 1 (D1) | 106.7 (33.1) | 94.4 (32.9)
  Day 5 (D5) | 114.5 (35.5) | 103.7 (28.0)

5. Secondary Outcome: Spatiotemporal Gait Characteristic (Step Length Symmetry - Symmetry Index)
Description: Step length [cm] of the weaker and stronger limbs were collected via instrumented walkway (GAITRite, CIR Systems Inc., NJ, USA) as participants completed three, 10-Meter Walk Test trials at each time point. Average step length of each lower limb for each walk trial was computed from data obtained from the GAITRite system. Lower limbs were classified as stronger or weaker according to manual muscle test scores collected at baseline (D1). The average step length for the stronger and weaker limbs was used to calculate the step symmetry index (SI) using the following formula: SI = ((SLs - SLw)/0.5(SLs + SLw)) x 100; where SLs = stronger limb stride length and SLw = weaker limb stride length. Final values are reported as the absolute % of the ratio difference in step length between the stronger and weaker limbs. A SI value of 0% indicates perfect interlimb step symmetry. Higher SI values indicate greater interlimb step length asymmetry.
Time Frame: D1, D5
Measure: Mean (Standard Deviation); unit: Absolute % of step length diff ratio
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
Absolute % of step length diff ratio
  Day 1 (D1) | 14.6 (12.2) | 12.3 (7.4)
  Day 5 (D5) | 16.2 (20.8) | 13.6 (11.8)

6. Secondary Outcome: Maximal Isometric Dorsiflexor Strength
Description: Ankle dorsiflexion (tibialis anterior) strength was measured with the subject seated and with the test foot strapped to a handheld dynamometer. An ankle dorsiflexion test was selected based on evidence indicating that the tibialis anterior is under the greatest corticospinal control. Maximum dorsiflexion force was calculated based on the highest force measured over three attempts. Results are reported for data obtained at baseline Day-1 (D1) and at follow-up on Day-5, 24-hours post-intervention.
Time Frame: D1, D5
Measure: Median (Inter-Quartile Range); unit: lbs
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
lbs
  Day 1 (D1) | 57.7 [34.4 to 72.8] | 68.3 [57.3 to 82.0]
  Day 5 (D5) | 49.3 [31.8 to 64.5] | 72.9 [57.6 to 92.9]

7. Secondary Outcome: Berg Balance Scale
Description: Balance was measured using the Berg Balance Scale (BBS), which has been found to be valid for use in persons with SCI. The BBS total score was calculated for each participant at each time point, and the median score for each group was calculated. The total range of scores for the BBS equals 0-56, with higher scores from baseline indicating greater balance performance and lower scores from baseline indicating worsened balance performance. Data reported were obtained at baseline Day-1 (D1) and at follow-up on Day-5, 24-hours post-intervention.
Time Frame: D1, D5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
score on a scale
  Day 1 (D1) | 38.0 [25.5 to 50.8] | 46.0 [39.0 to 51.0]
  Day 5 (D5) | 41.5 [29.3 to 46.8] | 49.0 [39.5 to 54.0]

8. Secondary Outcome: Falls Efficacy Scale-International Version (FES-I)
Description: The fear of falling may be a major concern for persons with mobility impairments and may limit one's confidence or ability to perform activities of daily living. Fear of falling may also limit an individual's performance of specific overground motor tasks irrespective of functional ability to perform that task. Therefore, the fear of falling was an important factor to consider relative to the mobility interventions employed in the present study. The FES-I total score was calculated for each participant at each time point, and the median for each group was recorded. The total range of scores possible for the FES-I is equal to 16-64, with lower total scores indicating decreased fear of falling. Data reported were obtained at baseline Day-1 (D1) and at follow-up on Day-5, 24-hours post-intervention.
Time Frame: D1, D5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
score on a scale
  Day 1 (D1) | 34.0 [29.3 to 40.0] | 33.0 [30.5 to 43.5]
  Day 5 (D5) | 33.5 [28.5 to 36.8] | 28.0 [26.0 to 43.5]

9. Secondary Outcome: Spinal Cord Assessment Tool for Spastic Reflexes
Description: The Spinal Cord Assessment Tool for Spastic Reflexes (SCATS) was used to assess the impact of motor skill training + sham stimulation and motor training + tDCS on spasticity. SCATS is well correlated with electrophysiological measures of spasticity and is better correlated with self-reported measures of spasm frequency than the Ashworth test. Total SCATS scores for each limb were summed and median values were obtained for each group. The total range of scores possible for the SCATS is 0-18, with a total score of 0 indicating no lower limb spasticity and higher total scores indicating greater spasticity severity. Data reported were obtained at baseline Day-1 (D1) and at follow-up on Day-5, 24-hours post-intervention.
Time Frame: D1, D5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
score on a scale
  Day 1 (D1) | 4.0 [2.0 to 7.5] | 4.0 [2.0 to 6.5]
  Day 5 (D5) | 6.0 [3.5 to 7.0] | 4.0 [1.0 to 7.0]

10. Secondary Outcome: Modified 5-Times Sit-to-Stand
Description: The modified 5-times sit-to-stand test was used as a measure of functional lower extremity strength. In this test, the participant was seated on a mat table with height adjusted to 80% of lower extremity length. The time required to complete 5 repetitions of standing up and sitting down (without using the upper extremities for assistance) was recorded. The average time to complete the test was calculated at each time point for each group. Lower sit-to-stand times indicate greater functional lower extremity strength. Results are reported for data obtained at baseline Day-1 (D1) and at follow-up on Day-5, 24-hours post-intervention.
Time Frame: D1, D5
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
seconds
  Day 1 (D1) | 13.7 (5.2) | 21.9 (17.3)
  Day 5 (D5) | 14.9 (7.3) | 19.6 (15.8)

11. Secondary Outcome: Maximal Isometric Quadriceps Strength
Description: Knee extensor (quadriceps) strength was measured with participants seated, with the test leg strapped to a handheld dynamometer. Prior studies have shown that a single session of tDCS improves quadriceps strength in persons with stroke. Maximum knee extensor force was analyzed based on the maximum force produced over three attempts. Results are reported for data obtained at baseline Day-1 (D1) and at follow-up on Day-5, 24-hours post-intervention.
Time Frame: D1, D5
Measure: Median (Inter-Quartile Range); unit: lbs
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
lbs
  Day 1 (D1) | 86.7 [63.6 to 114.3] | 92.1 [78.5 to 118.1]
  Day 5 (D5) | 84.4 [52.5 to 90.4] | 103.5 [85.4 to 131.9]

12. Secondary Outcome: 2 Minute Walk Test
Description: Functional walking capacity was measured based on 2-minute walk test distance. The use of the 2-minute rather than the 6-minute walk test allowed us to include individuals whose impairments result in inability to walk for 6 minutes. Total distance walked in 2-minutes was recorded for each participant at each time point, and the average distance was calculated for each group. Results are reported for data obtained at baseline Day-1 (D1) and at follow-up on Day-5, 24-hours post-intervention.
Time Frame: D1, D5
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
Number analyzed (Participants) | 14 | 11
m
  Day 1 (D1) | 83.1 (49.4) | 77.1 (55.3)
  Day 5 (D5) | 93.7 (50.3) | 86.7 (50.7)

ADVERSE EVENTS:
Time Frame: Adverse event queries and documentation were performed for each participant beginning at baseline on Day 1 and concluding following the last day of data collection on Day 5, which is the time course over which participants were enrolled in the study.
Groups:
- Motor Skill Training + Sham tDCS (MST+Sham-tDCS): Individuals will participate in 3 consecutive sessions of lower extremity motor skill training while receiving sham transcranial direct current stimulation (MST+sham-tDCS).
  MST: Motor skill training will consist of activities that will be performed while standing to promote upright control (the toe-tapping activity will be performed while seated). Participants will perform each of the 6 different activities for one minute each, until 4 cycles of the circuit have been completed (approximately 25 minutes total). Motor training activities will be performed at an intensity of 40-59% of heart rate reserve (HRR). Toe tapping will provide the opportunity for scheduled rest. During MST, all participants will wear a heart rate monitor to ensure that the optimal HR range is achieved. HRR will be calculated from resting and peak heart rate measures obtained during baseline testing via administration of a graded-exercise test.
Arm/Group | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) | Motor Skill Training + tDCS (MST+tDCS)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 2/14 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motor Skill Training + Sham tDCS (MST+Sham-tDCS) (N=14) | Motor Skill Training + tDCS (MST+tDCS) (N=11)
Mild Headache (General disorders) | 0 (0) | 3 (3) — 3 participants experienced mild headache following stimulation.
Moderate Headache (General disorders) | 1 (1) | 0 (0) — 1 participant reported a moderate headache following intervention.
Muscle Soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — 2 participants experienced muscle soreness following motor training.
Suprapubic Catheter Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — 1 participant reported skin irritation following motor training.
Thumb Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — 1 participant developed a blister on the thumb from holding on to a fixed bar during motor training.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT03237234/Prot_SAP_001.pdf